CLINICAL TRIAL: NCT04368312
Title: Psychological Impairment Due to Covid-19 in Hospital Staff
Brief Title: Psychological Impairment Due to Covid-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: TEMP553914-BO
Record Dates: First submitted 2020-04-09; First posted 2020-04-29 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Psychological Distress; Quality of Life
Keywords: quality of life; psychological distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health care providers/hospital staff: The targeted group are doctors and nurses (hospital stuff) of a large university hospital directly confronted with patients with Cov-19
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, just of questionnaire including validated tests

SUMMARY:
Hospital staff and emergency personnel are expected to suffer impaired psychological outcomes during a pandemic in terms of Quality of Life, anxiety, depression or other outcomes. The Covid-19 pandemic is a threat for both somatic and psychological health, therefore the impact of the impairment of this event on psychological parameters has to be assessed.

DETAILED DESCRIPTION:
Hospital staff and emergency personell are confronted with severe and life-threatening situations, therefore this group is considered to be at risk for impaired psychological health. A pandemic such as the Covid-19 endemic is suggested to severely impair the psychological state of this profession, amongst others Quality of life, anxiety, depression and other parameters. Therefore, it is crucial to assess the impact of impairment due to this global threat on the psychological health of health care providers. We therefore designed this study to evaluate baseline psychological characteristics and to re-assess those values in an interval of 60 days.

ELIGIBILITY:
Inclusion Criteria:

Hospital staff (doctors and nurses)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of all persons which can be attributed to hospital stuff, those include doctors and nurses (male/female)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
PCL5 Questionnaire | 14 days
  Validated 20-items questionnaire for PTSD
BSI - Brief symptom inventory | 14 days
  The Brief Symptom Inventory (BSI) is a 53-item screener for mental health problems with 9 subscales.
PHQD | 14 days
  Instrument for psychological diagnostics, able to test the severity of mental disorders and the success of their treatment
WHO - QoL BREF | 14 days
  Qol Questionnaire, assessed QoL with respect to the individual's perceptions in the context of culture and value systems.
STAXI | 14 days
  The State-Trait Anger Expression Inventory is used to measure the expressions & control of anger
AUDIT questionnaire | 14 days
  The AUDIT questionnaire is designed to help in the self assessment of alcohol consumption

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wesemann U, Hadjamu N, Wakili R, Willmund G, Vogel J, Rassaf T, Siebermair J. Gender Differences in Anger Among Hospital Medical Staff Exposed to Patients with COVID-19. Health Equity. 2021 Apr 19;5(1):181-184. doi: 10.1089/heq.2020.0119. eCollection 2021. PMID 33937603